CLINICAL TRIAL: NCT01420471
Title: Medicated Punctured-Glove-Finger Spacer Study
Acronym: FISHNET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, MD, FRCSC FARS, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FISHNET-2011
Record Dates: First submitted 2011-08-18; First posted 2011-08-19 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Sinusitis
Keywords: Endoscopic Sinus Surgery; Triamcinolone; Merocel Middle Meatus Spacers
MeSH Terms: conditions — Sinusitis | interventions — Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline-impregnated spacer (Active Comparator): Saline-impregnated spacers are actively being used as the standard of care. It does not contain any active ingredients.
  Interventions: Other: Saline-impregnated spacer
- Triamcinolone-impregnated spacer (Experimental): This study arm receives the experimental treatment, a Triamcinolone-impregnated spacer.
  Interventions: Drug: Triamcinolone

INTERVENTIONS:
Drug: Triamcinolone — Spacer will be impregnated with 2mL of Triamcinolone. The triamcinolone-impregnated spacer will be inserted into the middle meatal space after surgery. The spacer will be left in the middle meatus for a period of 6 days following surgery.
  Other Names: Triamcinolone-impregnated Middle Meatus Spacer; Experimental treatment; Endoscopic Sinus Surgery
  Arms: Triamcinolone-impregnated spacer
Other: Saline-impregnated spacer — Spacer will be impregnated with 2mL of Saline solution. The saline-impregnated spacer will be inserted into the middle meatal space intraoperatively. The spacer will be left in the middle meatus for a period of 6 days following surgery.
  Other Names: Saline-impregnated middle meatal spacer; Endoscopic sinus surgery; Control
  Arms: Saline-impregnated spacer

SUMMARY:
All adult patients undergoing sinus surgery for chronic rhinosinusitis (CRS) that satisfy the inclusion/exclusion criteria will be included in the study.

All patients enrolled in this study will have spacers (impregnated with saline or Triamcinolone) inserted into their middle meati after sinus surgery. Patients will serve as their own controls. Nostril's will be randomized to either the experimental treatment (Triamcinolone-impregnated spacer) or the control treatment (Saline-impregnated spacer). These spacers will be removed after 6-days post-op.

Participants will undergo the standard post-operative endoscopic sinus surgery follow-up appointments plus one additional research visit (not standard of care). This includes follow-up appointments at 6 days, 14 days, 5 weeks, 3 months, and 6 months of the post-operative period. During these appointments, the surgeon will assess the post-operative mucosal appearance (Philpott-Javer Sinus Rating System). SNOT-22 surveys will be administered, as per standard protocol, at each post-op follow up visit.

Sinus tissue biopsies will be taken from both meati on 28-day and 3-month post-op follow-up appointments for analysis.

Our objective is to determine if triamcinolone soaked Merocel middle meatus spacers (MMS) in a perforated glove finger improves patient outcomes, wound healing and reduces inflammation compared to a standard saline-soaked merocel sponge within a perforated glove finger in CRS patients receiving FESS.

Our hypothesis is that triamcinolone-medicated Merocel MMS are not inferior to standard saline-soaked spacers, when both are enclosed in a perforated surgical glove finger.

DETAILED DESCRIPTION:
Patients suffering from chronic rhinosinusitis undergoing Functional Endoscopic Sinus Surgery (FESS) require nasal spacers to be inserted intra-operatively into the middle-meatus to prevent lateralization of the middle turbinate and subsequent scarring and adhesions. Nasal spacers can be impregnated with topical steroids to assist in post-surgical recovery. Our centre is now investigating the effect of triamcinolone-medicated nasal spacers placed inside a punctured glove finger to improve wound healing.

All patients enrolled in this study will have spacers (impregnated with saline or Triamcinolone) inserted into their middle meati after sinus surgery. Patients will serve as their own controls. One nostril will receive the experimental treatment (Triamcinolone-impregnated spacer) and one will receive the control treatment (Saline-impregnated spacer). These spacers will be removed after 6-days post-op.

Randomization of patients' nostrils to a treatment arm will occur on the day of surgery based on a closed envelope system.

Participants will undergo the standard post-operative endoscopic sinus surgery follow-up appointments plus one additional research visit (not standard of care). This includes follow-up appointments at 6 days, 14 days, 5 weeks, 3 months, and 6 months of the post-operative period. The 14-day follow-up appointment is an additional visit not included as standard practice at our centre. However, study patients will have this added visit in order to closely observe their recovery and endoscopic evaluation. During these appointments, the surgeon will assess the post-operative appearance (Philpott-Javer Sinus Rating System), number of infections, pain, and 1st week post-operative bleeding (only at 6 day visit).

The Sino-Nasal Outcome Test (SNOT-22) questionnaire is to be completed by the study participants at 6 days, 14 days, 5 weeks, and 3 months of the post-operative period. The SNOT-22 is a 5-minute questionnaire consisting of 22 questions, which asks participants to rate their sinus symptoms and social/emotional consequences of their nasal disorder from "no problem" to "problem as bad as it can be."

Sinus tissue biopsies will also be taken from both meati intraoperatively (standard of care) and on 28-day and 3-month post-op follow-up appointments (above standard of care). Biopsies will be sent to a pathologist for grading on a scale of tissue inflammation. To grade the level of mucosal inflammation in an objective fashion, the pathologist has previously devised a grading system on a scale from 0 to 4. A score of 0 is given for normal tissue, 1 for submucosal inflammation with no inflammatory infiltrate into the epithelium, 2 for inflammatory infiltrate with neutrophils into the epithelium with no evidence of necrosis, 3 for inflammatory infiltrate with neutrophils into the epithelium with evidence of focal necrosis and 4 for inflammatory infiltrate with neutrophils into the epithelium with evidence of extensive necrosis (5).

ELIGIBILITY:
Inclusion Criteria:

* All CRS patients undergoing bilateral endoscopic surgery requiring spacers

Exclusion Criteria:

* Patients under the age of 19
* Patients unable to understand English
* Patients who are pregnant
* Patients with known bleeding disorders
* Patients with systemic disorders affecting the nose
* Patients in another concurrent study
* Unilateral endoscopic sinus surgery
* Surgery in which spacers are not needed
* Patients undergoing sinonasal tumour resection
* Patients who cannot tolerate or are allergic to triamcinolone

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Post-operative endoscopic appearance | Participants will be followed for the duration of post op standard of care, an expected average of 6 months.
  Participants in the study have their sinus cavities assessed by rigid endoscopy and mucosa graded by the Lund-Kennedy and Philpott-Javer scaling system. Each sinus cavity (frontal, ethmoid, maxillary and sphenoid) and olfactory cleft will be given a score between zero and nine, with an extra point for the presence of fungal mucin, achieving a total potential maximum out of fifty per side (14).
Post-operative inflammation | Biopsies will be removed during a 3 month period (beginning the day of surgery)
  Participants will have biopsies taken from both middle meati in contact with nasal packing. Biopsies will be assessed and scored with a previously utilized histologic scoring system at our centre in order to determine the level of inflammation between the triamcinolone-medicated and saline-soaked spacers.

SECONDARY OUTCOMES:
Post-Operative SNOT-22 | Participants will be followed for the duration of post op standard of care, an expected average of 6 months.
  Sino-Nasal Outcome Test (SNOT-22) is current standard in Rhinology for the assessment of the patient's subjective sinus symptoms and its effect on their daily functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Amin R Javer, MD, FRCSC,FARS, Principal Investigator — St. Paul's Hospital, Canada
Locations (1):
- E.N.T. Clinic, St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Desrosiers M, Hussain A, Frenkiel S, Kilty S, Marsan J, Witterick I, Wright E. Intranasal corticosteroid use is associated with lower rates of bacterial recovery in chronic rhinosinusitis. Otolaryngol Head Neck Surg. 2007 Apr;136(4):605-9. doi: 10.1016/j.otohns.2006.10.028. PMID 17418259
- [Result] Chang EH, Alandejani T, Akbari E, Ostry A, Javer A. Double-blinded, randomized, controlled trial of medicated versus nonmedicated merocel sponges for functional endoscopic sinus surgery. J Otolaryngol Head Neck Surg. 2011 Feb;40 Suppl 1:S14-9. PMID 21453656
- [Result] Shoman N, Gheriani H, Flamer D, Javer A. Prospective, double-blind, randomized trial evaluating patient satisfaction, bleeding, and wound healing using biodegradable synthetic polyurethane foam (NasoPore) as a middle meatal spacer in functional endoscopic sinus surgery. J Otolaryngol Head Neck Surg. 2009 Feb;38(1):112-8. PMID 19344620
- [Result] Franklin JH, Wright ED. Randomized, controlled, study of absorbable nasal packing on outcomes of surgical treatment of rhinosinusitis with polyposis. Am J Rhinol. 2007 Mar-Apr;21(2):214-7. doi: 10.2500/ajr.2007.21.3011. PMID 17424883